CLINICAL TRIAL: NCT04988178
Title: Retrospective Analysis of Naive Patients With Age-related Macular Degeneration Neovascular Type and Treated With Ranibizumab (Lucentis®) in Treat-and-extend at the CHU Brugmann.
Brief Title: Analysis of naïve Patients With Age-related Macular Degeneration Neovascular Type and Treated With Ranibizumab (Lucentis®) in Treat-and-extend at the CHU Brugmann.
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Laurence Postelmans, Head of ophtalmology department, Brugmann University Hospital
Other Study IDs: CHUB- KIERKOWICZ
Record Dates: First submitted 2021-05-10; First posted 2021-08-03 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Age-related macular degeneration (AMD) is a leading cause of blindness in people over 50 years old. Neovascular AMD, the most severe form and the most severe is characterized by the appearance, spread and growth of subretinal neovessels. One of the major molecular mediators is the endothelial growth factor vascular (VEGF).

Intra-vitreous (IVI) injection of an anti-VEGF may slow the progression of Neovascular AMD and stabilize vision in the majority of cases. Ranibizumab (Lucentis®) is one of the anti-VEGF molecules approved in Belgium to treat neovascular AMD.

At the start of its use, ranibizumab was first injected monthly and then according to the "reactive" protocol. Over time, a new strategy of treatment was born: the "treat-and-extend" (T&E). This is 'made to measure' protocol for each patient aiming to reduce the frequency of injections while guaranteeing inactivity of the disease. It starts with the loading dose, i.e. 3 injections given 4 weeks apart. Subsequently, the interval is lengthened by slices of 1 or 2 weeks provided that the visual and anatomical results remain stable. In the event of deterioration, the interval is shortened while keeping a minimum of 4 weeks between each IIV.

The efficacy and safety of ranibizumab, when used in a proactive regimen of T&E, has been shown in the CANTREAT randomized controlled trial. However, there is a lack of more data on T&E used in current practice, and particularly on the number of injections and treatment intervals over a minimum treatment period of 24 months.

The aim of this retrospective study carried out at the CHU Brugmann Hospital is to determine the number of injections and the intervals necessary to have encouraging results in visual acuity over a treatment period of at least two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 50 years old diagnosed with neovascular age related macular degeneration,
* Patients who have never received anti-VEGF treatment,
* Patients who started intra-vitreous injections of ranibizumab between 01 January 2014 and November 30, 2019,
* Treatment by "treat-and-extend" directly after the loading dose of ranibizumab,
* Availability of the medical file reporting treatment with ranibizumab.

Exclusion Criteria:

* Participation in an interventional clinical study during treatment with ranibizumab,
* Patients suffering from ocular pathologies and having required surgery during the first 24 months of treatment with ranibizumab (for example advanced glaucoma or cataract).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Naive patients with age-related macular degeneration, neovascular type, treated with ranibizumab (Lucentis®) in "treat-and-extend" at the CHU Brugmann Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Injections number (first 24 months of treatment) | first 24 months of treatment
  Number of injections during the first 24 months of treatment
Injections interval | during the 2nd year of treatment
  Last injection interval during the 2nd year of treatment, in weeks

SECONDARY OUTCOMES:
Injection number (up to 4 years of treatment) | up to 4 years of treatment
  Number of injections during the 1st, 2nd, 3rd and 4th year of treatment
Injections interval (up to 4 years of treatment) | up to 4 years of treatment
  Last injection interval during the 1st, 2nd, 3rd and 4th year of treatment (if applicable), in weeks
Most stable injection interval | up to 4 years of treatment
  Most stable injection interval during the 2nd, 3rd and 4th year of treatment (if applicable), in weeks
Overall extension interval | up to 4 years of treatment
  Expected overall extension interval: by 1 week, 2 weeks, 3 weeks or 4 weeks
Covid 19 impact | up to 4 years of treatment
  Impact of Covid-19 on the injection interval
Number of follow-up visits | up to 4 years of treatment
  Number of follow-up visits during each year of treatment
Visual acuity | up to 4 years of treatment
  Visual acuity at baseline, after 90 days and at the end of each year of treatment in the study
Age | Baseline
  Age of the patient at baseline
Eye lesion type | Baseline
  Eye lesion type
Fluid | Baseline
  Presence or absence of intra-retinal fluid, subretinal fluid, detachment of the pigment epithelium
Fluid | 90 days after baseline
  Presence or absence of intra-retinal fluid, subretinal fluid, detachment of the pigment epithelium
Fluid | once a year up to 4 years of treatment
  Presence or absence of intra-retinal fluid, subretinal fluid, detachment of the pigment epithelium
Date of first symptoms | Baseline
  Date of first symptoms of neovascular AMD
Date of first injection | Baseline
  Date of first ranibizumab injection
Retinal thickness | up to 4 years of treatment
  Retinal thickness at baseline, after 90 days and at the end of each year of treatment
Treatment regimen | first 12 months of treatment]
  Has there been a change in treatment regimen after the first 12 months of treatment?
Number of patients stopping treatment (12-24 months) | between 12 and 24 months of treatment
  Number of patients stopping treatment between 12 and 24 months of treatment
Reason for stopping treatment (12-24 months) | between 12 and 24 months of treatment
  Reason for stopping treatment between 12 and 24 months of treatment
Number of patients stopping treatment (24-36 months) | between 24 and 36 months of treatment
  Number of patients stopping treatment between 24 and 36 months of treatment
Reason for stopping treatment (24-36 months) | between 24 and 36 months of treatment
  Reason for stopping treatment between 24 and 36 months of treatment
Number of patients stopping treatment (36-48 months) | between 36 and 48 months of treatment
  Number of patients stopping treatment between 36 and 48 months of treatment
Reason for stopping treatment (36-48 months) | between 36 and 48 months of treatment
  Reason for stopping treatment between 36 and 48 months of treatment
Number of patients stopping treatment (first 12 months) | First 12 months of treatment
  Number of patients who stopped treatment in the first 12 months
Reason for stopping treatment (first 12 months) | First 12 months of treatment
  Reason for stopping treatment in the first 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Postelmans, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No